**Study Title**: Randomized controlled trial to test the feasibility, acceptability, and preliminary effectiveness of a psychosocial intervention to support Alzheimer's family caregivers in Vietnam.

**NCT#**: NCT03587974

Document Date: March 1, 2020

**Document Type**: Statistical Analysis Plan

## Statistical Analysis Plan

Characteristics of the caregivers and the care recipients will be compared between the two groups using a two-sample t-test or Chi-square test; the Wilcoxon rank sum test or Fisher's exact test will be used if needed due to violations of the underlying assumptions. Primary analysis of the intervention effect will use an intent-to-treat approach, in which groups were compared based on randomization assignment. To account for the clustering of participants by commune, mixed effects models that included a cluster-specific random effect will be used to estimate differences between groups. Models will utilize the post-intervention assessment as the outcome and included the baseline assessment as a covariate. The post-intervention assessment will be divided by the standard deviation in the entire sample at baseline, so that interpretation of model coefficients will be in terms of standard deviation units. Model assumptions will be checked and met by the data. All analyses will be conducted in SAS, version 9.4, and a *p*-value less than 0.05 considered statistically significant.